CLINICAL TRIAL: NCT06635421
Title: The Expand Study-Pharmacist Administered Long Acting Cabotegravir + Rilpivirine to Expand Access for People With HIV
Acronym: EXPAND
Status: Not yet recruiting | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Corrilynn Hileman, Medical Director of the Infectious Disease Clinic, Associate Professor of Medicine, MetroHealth Medical Center
Other Study IDs: STUDY00000459
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: HIV I Infection
Keywords: long acting injectable antiretroviral therapy; cabotegravir; rilpivirine; HIV; pharmacist administered medication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient participants receiving in clinic nurse administered long-acting injectable ART: People with HIV on long acting cabotegravir + rilpivirine who elect to continue to receive their injections in clinic by a nurse
  Interventions: Other: Model of care delivery for long-acting injectable ART
- Patient participants receiving pharmacist administered long-acting injectable ART in pharmacy: People with HIV on long acting cabotegravir + rilpivirine who elect to continue to receive their injections in a satellite pharmacy by a pharmacist
  Interventions: Other: Model of care delivery for long-acting injectable ART
- Staff participants: Staff involved in the long-acting injectable ART workflow

INTERVENTIONS:
Other: Model of care delivery for long-acting injectable ART — This study is assessing a novel model of care delivery, i.e. pharmacist administered long-acting cabotegravir + rilpivirine (CAB+RPV LA). In phase 2 and 3, no medication will be provided by the study. The decision to initiate CAB+RPV LA will be at the discretion of the patient and their provider in accordance with both standard of care and local prescribing practices. This will occur independent of study participation. The study intervention is the model of care for CAB+RPV LA administration. The models of care being studied include (1) pharmacist administered CAB+RPV LA in MetroHealth satellite pharmacy setting (novel model of care); (2) nurse administered CAB+RPV LA in the Infectious Diseases clinic at MetroHealth main campus (current standard of care).
  Groups: Patient participants receiving in clinic nurse administered long-acting injectable ART; Patient participants receiving pharmacist administered long-acting injectable ART in pharmacy

SUMMARY:
The purpose of The EXPAND study is to develop and pilot a pharmacist led model of medication delivery. Following a co-design phase, patients may receive injections at satellite pharmacies by a licensed pharmacist. The acceptability, appropriateness, and feasibility of this approach and standard in clinic administration by a nurse will be assessed.

DETAILED DESCRIPTION:
The EXPAND study will involve three phases:

Phase 1 A care delivery model incorporating pharmacist administered CAB+RPV LA at satellite pharmacies will be developed using codesign. A core group of stakeholders will be engaged in codesigning the intervention. Stakeholders will include HIV physicians, HIV nurses, electronic health record informatics experts, pharmacists, and 3 PWH who are currently receiving CAB+RPV LA. Engaging with patients in codesign ensures patient experience and input is incorporated since the primary goal is improving their health. Bringing stakeholders together to generate solutions ahead of the implementation significantly impacts buy-in.

Codesign team meetings will be convened as hybrid one hour meetings, i.e., in person with option for attendance via virtual platform - Webex or Zoom. There will be 5-6 design team meetings. Number of meetings will depend on progress towards producing a process map outlining the pharmacist administered CAB+RPV LA model of care. Content of meetings will include: introduction to codesign and EXPAND; establishment of current workflow for CAB+RPV LA administration by nurse in clinic; determination of essential components; production of process map outlining pharmacist administered CAB+RPV LA work flow; outlining changes from prior work flow to inform clinical staff education, make changes to electronic health record tools. The final process map will be sent to design team members for verification and additional recommendations.

After the design team work is complete, semi-structured interviews with design team members will be conducted to evaluate the codesign process to improve codesign internally and disseminate findings to inform best practices for conducting codesign activities for models of HIV care delivery and treatment for HIV. These interviews will be performed by trained interviewers from the Population Health Institute at MH. Interviews will take place by phone or in a private room, and audio recordings will later be transcribed verbatim.

Phase 2 After completion of codesign process, a single arm, pilot study of the pharmacist administered CAB+RPV LA model will be performed at a pilot site. Four patient participants with diverse backgrounds will be enrolled and all will receive their CAB+RPV LA in the pharmacist administered CAB+RPV LA model. After 1 dose of CAB+RPV LA are administered by a pharmacist at a satellite MetroHealth pharmacy, semi-structured in-depth qualitative interviews with each participant, pharmacist, and nurse post-pilot will inform the final pharmacist administered CAB+RPV LA model.

Guided by the Consolidated Framework for Implementation Research (CFIR), these initial qualitative interviews will focus on illuminating insight to participants' (i.e., innovation recipients') impressions of, specifically, the innovation relative advantage (e.g., benefits and quality of the pharmacist-administered CAB+RPV LA model compared to current practice) and innovation adaptability (e.g., how participants' experience of receiving pharmacist-administered injections aligns with their own and peers' needs). These interviews will be performed by trained interviewers from the Population Health Institute at MH. Interviews will take place in a private room, and audio recordings will later be transcribed verbatim. This data will be aggregated and utilized to refine the intervention toward maximally appropriate design, complexity, and usability for Phase 3.

Phase 3 Finally, a parallel arm, 48-week, prospective, non-randomized study of the pharmacist administered CAB+RPV LA model and the in clinic nurse administered CAB+RPV LA model will be completed. Both patient (N=140) and staff (N=20) participants will be enrolled and a mixed methods approach will be performed. The decision to initiate CAB+RPV LA is at the discretion of the patient and their provider, i.e. study staff will not participate in this decision.

The Proctor Framework will be used to evaluate implementation outcomes focusing on acceptability, appropriateness, and feasibility. All participants (patients and staff) will complete the previously validated Acceptability of Intervention Measure (AIM) and Intervention Appropriateness Measure (IAM), and staff participants also complete the Feasibility of Intervention Measure (FIM) at baseline, week 16 and 48. CFIR will comprehensively guide semi-structured qualitative interviews to complement the structured surveys and develop a more nuanced understanding of patient and staff perspectives of the novel pharmacist administered CAB+RPV LA model. Interviews of a subset of patient participants will occur at baseline, and 48 weeks. In-depth interview guides will be developed to inquire along specific CFIR domains of innovation (e.g., how calibrated is the pharmacist-administered innovative treatment to patients' clinical and psychosocial needs?), inner setting (e.g., how do physical and relational infrastructure components of the treatment setting support patients' treatment and wellbeing?), and individuals (e.g., how do patients as innovation recipients view treatment innovations as aligning with their own priorities, preferences, and needs?). Interviews of all staff participants will occur 48 weeks after the initial patient participant is enrolled and will focus on facilitators and barriers to sustainability. Interviews will be performed by trained interviewers from the Population Health Department at MH throughout the study. These interviews will take place in a private room, and audio recordings will later be transcribed verbatim.

Approach to participants who switch groups during study: Participants who decide to switch to the other model of care after the entry visit will be allowed to continue on study. Week of switch will be captured. Each switch participant will be approached for qualitative interview to assess reasons for switch. Data will continue to be collected as per schedule of evaluations.

ELIGIBILITY:
Patient Participant Inclusion Criteria:

* 18 years of age and older
* diagnosed with HIV by approved HIV screen and confirmation test
* currently on CAB+RPV LA every 4 or 8 weeks
* has received at least two doses of CAB+PRV LA
* last HIV-1 RNA <50 copies/ml
* no known or suspected resistance to either cabotegravir or rilpivirine
* no plans to change medication in the next 48 weeks
* no plans to move out of state
* has plans to avoid pregnancy if of reproductive potential

Patient Participant Exclusion Criteria:

* individuals who are unable or unwilling to adhere to the study protocol
* unable to speak/comprehend English
* insurance coverage for medication through medical benefit

Staff Participant Inclusion/Exclusion Criteria:

-all available staff involved in the CAB+RPV LA workflow will be approached for inclusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient participants will be recruited from the MetroHealth System's HIV provider clinics. Any patient who has decided with their provider to initiate CAB+RPV LA and has received at least two doses of CAB+RPV LA through in clinic nurse administration will be considered for enrollment. Decision to initiate CAB+RPV LA is made by a treating HIV physician with their patient and then is reviewed by an HIV pharmacist. This occurs within the context of clinical care without involvement of the study investigators. Staff participants will be recruited from nursing and physician staff in the HIV clinic, and pharmacy staff at the MetroHealth satellite pharmacies.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of intervention | Entry, Week 16, Week 48
  Acceptability of Intervention Measure (AIM)
Intervention appropriateness | Entry, Week 16, Week 48
  Intervention Appropriateness Measure (IAM)
Feasibility of Intervention | Entry, Week 16, Week 48
  Feasibility of Intervention Measure (FIM) completed by staff participants only

SECONDARY OUTCOMES:
Facilitators and barriers to model of care | Entry, Week 48
  Semi-structured interviews conducted with patient participants
Organizational facilitators and barriers to sustainability for model of care | Week 48
  Semi-structured interviews conducted with staff participants
Fidelity | Week 16, Week 48
  Proportion of CAB+RPV LA doses entry given within manufacturer's recommended dosing window
Fidelity | Entry, Week 16, Week 48
  Length of injection visits in minutes
HIV treatment satisfaction | Entry, Week 16, Week 48
  HIVTSQs
HIV treatment satisfaction | Week 48
  HIVTSQc
Quality of life | Entry, Week 48
  36-Item Short Form Survey
HIV stigma | Entry, Week 48
  HIV stigma survey
Virologic suppression | Week 16, Week 48
  Proportion with HIV-1 RNA <=20
Confirmed virologic failure | Week 16, Week 48
  2 consecutive HIV-1 RNA >=200
Treatment emergent resistance | Week 16, Week 48
  Incidence of treatment emergent resistance
Adverse events | Week 16, Week 48
  Incidence and severity of adverse events
Participant discontinuation | Week 16, Week 48
  Proportion of patient participant discontinuation due to adverse events, incidence and severity of injection site reactions
Injection site reactions | Entry, Week 16, Week 48
  Incidence and severity of injection site reactions
Engagement in HIV care | Week 48
  Proportion of HIV provider visits attended
Missed HIV provider appointments | Week 48
  Proportion of no shows to HIV provider visits
Routine HIV lab completion | Week 48
  Proportion with routine HIV labs done
Routine cholesterol lab completion | Week 48
  Proportion with routine cholesterol done
Routine renal function lab completion | Week 48
  Proportion with routine renal function lab done - serum creatinine or urine protein
Routine blood glucose assessment completion | Week 48
  Proportion with routine blood glucose assessment done - fasting blood glucose or hemoglobin A1C
Routine sexually transmitted infection screening completion | Week 48
  Proportion with routine screening for sexually transmitted infections - urine, or throat, or rectal gonorrhea, chlamydia, trichomonas screen, or syphilis serology in blood

CONTACTS AND LOCATIONS:
Overall Officials: Corrilynn O Hileman, MD, Principal Investigator — MetroHealth System, Ohio

IPD SHARING:
Plan to Share IPD: No
To collaborate regarding data collected as part of this study, please contact the PI.